CLINICAL TRIAL: NCT06036589
Title: Characterization of Bovine Adrenal Medulla (BAM8-22) as a New Surrogate Model of Non-histaminergic Itch
Brief Title: Characterization of Bovine Adrenal Medulla as a Model of Non-histaminergic Itch
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Giulia Erica Aliotta, Principal Investigator, PhD fellow, Aalborg University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Basic Science
Other Study IDs: N-20190062 3rd project
Record Dates: First submitted 2022-03-09; First posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Itch
MeSH Terms: conditions — Pruritus | interventions — bovine adrenal medulla 8-22

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CA application + BAM8-22 (Experimental)
  Interventions: Drug: CA and BAM8-22; Drug: Vehicle and BAM8-22 application
- CA application and vehicle (Experimental)
  Interventions: Drug: CA; Drug: vehicle

INTERVENTIONS:
Drug: CA and BAM8-22 — CA (tran-cinnamaldheyde) solution (in ethanol 5%) application and BAM8-22 with inactivate cowhage spicules 20 µl of BAM8-22 will be applied to a previously determined area on the volar forearm using inactivate cowhage spicules
  Arms: CA application + BAM8-22
Drug: Vehicle and BAM8-22 application — Vehicle (ethanol) application and BAM8-22 with inactivate cowhage spicules 20 µl of BAM8-22 will be applied to a previously determined area on the volar forearm using inactivate cowhage spicules
  Arms: CA application + BAM8-22
Drug: CA — CA (tran-cinnamaldheyde) solution (in ethanol 5%) application to a previously determined area on the volar forearm
  Arms: CA application and vehicle
Drug: vehicle — Vehicle (ethanol) application and inactivate cowhage spicules will be applied to a previously determined area on the volar forearm
  Arms: CA application and vehicle

SUMMARY:
With this experiment, the experimenter wish evaluate the role of TRPA1 on non-histaminergic itch induced by BAM8-22

DETAILED DESCRIPTION:
With this experiment, the experimenter wish evaluate the role of TRPA1 on non-histaminergic itch induced by BAM8-22 2 (Bovine Adrenal Medulla), which is found naturally in the human body and which has proved to evoke itch. To evaluate the role of TRPA1 it will be used a TRPA1 agonist

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* 18-60 years
* Speak and understand English

Exclusion Criteria:

* Pregnancy or lactation
* Drug addiction defined as any use of cannabis, opioids or other drugs
* Previous or current history of neurological, dermatological, immunological musculoskeletal, cardiac disorder or mental illnesses that may affect the results (e.g. neuropathy, muscular pain in the upper extremities, etc.)
* Moles, wounds, scars or tattoos in the area to be treated or tested
* Lack of ability to cooperate •
* Current use of medications that may affect the trial such as antihistamines and pain killers.
* Skin diseases
* Consumption of alcohol or painkillers 24 hours before the study days and between these
* Acute or chronic pain
* Participation in other trials within 1 week of study entry (4 weeks in the case of pharmaceutical trials)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
superficial blood perfusion | change from baseline, up to 10 minutes after the application
  is measured by a speckle contrast imager (FLPI, Moor Instruments, England)
Warm Detection Threshold | change from baseline, up to 10 minutes after the application
  the tests for thermal sensation will all be performed using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device
Heat Pain threshold | change from baseline, up to 10 minutes after the application
  the tests for thermal sensation will all be performed using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device
Cold Detection Threshold | change from baseline, up to 10 minutes after the application
  the tests for thermal sensation will all be performed using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device
Cold Pain threshold | change from baseline, up to 10 minutes after the application
  the tests for thermal sensation will all be performed using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device
Pain supra-threshold heat Stimuli | change from baseline, up to 10 minutes after the application
  the tests for thermal sensation will all be performed using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device
hyperknesis | change from baseline, up to 10 minutes after the application
  measured by using a mildy pruritic, non-painful von Frey filaments of a predetermined intensity (5-30 milliNewton of force). participants will rate the itch sensation induced by stimuli with von Frey filaments on an numerical rating scale from 0 to 10
mechanical pain threshold | change from baseline, up to 10 minutes after the application
  is performed using a pin-prick set (Aalborg University). The set consists of 8 needles each having a diameter of 0,6 mm and different force applications. it will be determinate a threshold corresponding to the force of the pinprick (mN) from which participants start to feel pain
mechanical pain sensitivity | change from baseline, up to 10 minutes after the application
  is performed using a pin-prick set (Aalborg University). The set consists of 8 needles each having a diameter of 0,6 mm and different force applications
itch rating | change from baseline, up to 10 minutes after the application
  the subject will rate the itch for 10 minutes by using a visual analog scale (VAS) on a tablet. this scale goes from 0 to 100. 0 indicates "no itch" and 100 indicates "worst imaginable itch"

SECONDARY OUTCOMES:
pain rating | change from baseline, up to 10 minutes after the application
  the subject will rate the pain for 10 minutes by using a visual analog scale (VAS) on a tablet. this scale goes from 0 to 100. 0 indicates "no pain" and 100 indicates "worst imaginable pain

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University, Aalborg, Denmark